CLINICAL TRIAL: NCT05066542
Title: Leveraging Recreational Basketball to Increase Participation in the National Diabetes Prevention Program (NDPP) Among Adults Aged 18-44 Years at Kaiser Permanente Georgia
Brief Title: Recreational Basketball to Increase Participation in Diabetes Prevention
Acronym: DPPHoops
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Felipe Lobelo, Physician Program Director Epidemiology, Public Health and Preparedness, TSPMG, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KP1546327; KPR-SM-2020-01/1 (Other Grant/Funding Number: Kaiser Permanente and National Basketball Association)
Record Dates: First submitted 2021-09-08; First posted 2021-10-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; PreDiabetes
Keywords: Prediabetes; National Diabetes Prevention Program; Weight loss; Physical Activity; Basketball
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Weight Loss; Motor Activity | interventions — 4-nitro-3-dimethylaminopropiophenone

STUDY DESIGN:
Intervention Model Description: The study is interventional Efficacy trial for people at risk for type 2 diabetes. Participants will be randomized into the traditional DPP curriculum or DPP + basketball. Certified NDPP coaches will deliver the curriculum.The Traditional arm will receive the standard NDPP curriculum. The intervention arm will receive the NDPP curriculum and participate in group based exercise sessions. Both groups will submit weekly activity reports.
  Group evaluations are based on the percentage of participants achieving 5% weight loss at 12-months; self-reported dietary intake, physical activity and sleep time, HbA1c, fasting glucose, body composition, blood pressure, aerobic fitness, musculoskeletal fitness, quality of life, self-efficacy, motivation and depression symptoms at 12-months. Assessments will be conducted at baseline, 6 months, and at 12-months from study initiation. An additional 24-month measurement will be conducted to determine sustainability of program effects.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NDPP Standard of Care SOC (Active Comparator): Participants in this arm will participate in the traditional NDPP program delivered virtually by certified NDPP coaches. During Months 1-4 participants will attend a 60-minute virtually facilitated session of the NDPP curriculum. During Months 5-8, virtual NDPP curriculum sessions will be held every two weeks. During Months 9-12, participants will attend a monthly 60-minute NDPP curriculum session. Participants will submit a weekly weight report during the 12 month participation and will complete the ASA 24 hour food recall every 90 days.
  Interventions: Behavioral: NDPP Standard of Care SOC
- NDPP + Basketball (BB) (Experimental): Participants in this arm will participate in the traditional NDPP program delivered virtually by certified NDPP coaches along with virtual fitness sessions and in-person basketball sessions. During Months 1-4, participants will attend a 60-minute virtually facilitated session of the NDPP curriculum, followed by a 30-minute virtual fitness session. During that same week, participants will meet in person, for a 90-minute BB session. During Months 5-8, virtual NDPP curriculum sessions will be held every two weeks and there will no longer be a 30-minute online fitness session succeeding the session. During this same four-month period, 60-minute, in-person BB sessions will be held weekly. During Months 9-12, participants will attend a monthly 60-minute NDPP curriculum session and bi-weekly 60-minute in-person BB sessions. Participants will submit a weekly weight report during the 12 month participation and will complete the ASA 24 hour food recall every 90 days.
  Interventions: Behavioral: NDPP + Basketball (BB)

INTERVENTIONS:
Behavioral: NDPP + Basketball (BB) — DPP Hoops: Participants in this arm will participate in the traditional NDPP program delivered virtually by certified NDPP coaches along with virtual fitness sessions and in-person basketball sessions. During Months 1-4, participants will attend a 60-minute virtually facilitated session of the NDPP curriculum, followed by a 30- minute virtual fitness session. During that same week, participants will meet in person, for a 90-minute BB session. During Months 5-8, virtual NDPP curriculum sessions will be held every two weeks and there will no longer be a 30-minute online fitness session succeeding the session. During this same four-month period, 60-minute, in-person BB sessions will be held weekly. During Months 9-12, participants will attend a monthly 60-minute NDPP curriculum session and biweekly 60-minute in-person BB sessions. Participants will submit a weekly weight report during the 12 month participation and will complete the ASA 24 hour food recall every 90 days.
  Other Names: DPP Hoops
  Arms: NDPP + Basketball (BB)
Behavioral: NDPP Standard of Care SOC — DPP: Participants in this arm will participate in the traditional NDPP program delivered virtually by certified NDPP coaches. During Months 1-4 participants will attend a 60-minute virtually facilitated session of the NDPP curriculum. During Months 5-8, virtual NDPP curriculum sessions will be held every two weeks. During Months 9-12, participants will attend a monthly 60-minute NDPP curriculum session. Participants will submit a weekly weight report during the 12 month participation and will complete the ASA 24 hour food recall every 90 days.
  Other Names: NDPP; Diabetes Prevention Program DPP
  Arms: NDPP Standard of Care SOC

SUMMARY:
The purpose of this study is to assess the efficacy of adapting the National Diabetes Prevention Program (NDPP) to include recreational sports in effort to increase physical activity (PA) and promote lifestyle changes that can help reduce the risk of developing Type 2 Diabetes Mellitus. The hypothesis is that both the traditional NDPP and the NDPP+ Basketball will be considered feasible. The primary outcome is to assess whether the intervention (NDPP+BB) compared to the standard of care (NDPP only) will result in greater weight loss, lower A1c, and increased engagement in physical activity.

DETAILED DESCRIPTION:
The NDPP has successfully helped to reduce the rate of Type 2 Diabetes Mellitus (T2DM) through moderate weight loss and increased physical activity(PA). Kaiser Permanente Georgia (KPGA) members, identified as being at risk to develop type 2 diabetes will be recruited to participate in the intervention trial testing DPP vs. NDPP+ BB study arms. Participants will be randomized into 1 of 2 groups (traditional DPP curriculum or DPP + basketball).

The central objective of this project is to determine the feasibility of adapting the NDPP to include recreational basketball as an exercise component among KPGA population of overweight, pre-diabetic adults ages 18-44 using novel translational science approach and qualitative formative research tools. The secondary objective is to implement the adapted NDPP + BB program among a pre-diabetic KPGA adult members, 18-44 years living in Atlanta and determine post-program efficacy in achieving the desired 5 percent weight loss goal.

The objective is to contribute beneficial information to clinical and operational leaders across KP and beyond, as they consider approaches to improve overall participation rates in the NDPP, particularly for young and middle-aged adult members, leveraging interest in a popular recreational team-based sport such as BB. Longer-term, the goal is to reduce diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-44 years
* BMI >= 25 kg/m2
* Previous diagnosis of prediabetes as defined:
* HbA1c 5.7 to 6.4% at baseline
* Not engaged in high exercise levels (self-report of less than 300 minutes of exercise per week)
* Not engaged in other lifestyle intervention program in past 2 years
* Ability to read in English and provide informed consent
* Ability to walk unassisted for 30 minutes
* Ability to jump in place

Exclusion Criteria:

* Diabetes due to underlying conditions
* Type 1 Diabetes
* Type 2 Diabetes
* End Stage Renal Disease (ESRD)
* Myocardial Infarction within the last 12 months
* Cancer treatment
* Congestive Heart Disease
* Not currently pregnant
* Any history of seizures or uncontrolled neurologic or psychiatric condition that may interfere with the intervention plan

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Percent Weight Loss Efficacy | 12 months
  Compare percent of program participants achieving 5% or more weight loss between the DPP Standard of care group and the DPP+BB intervention group.

SECONDARY OUTCOMES:
Blood pressure | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean systolic and diastolic blood pressure (mm Hg)
HbA1c | 12 month
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean HbA1c (percent)
Aerobic Fitness | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean aerobic fitness (ml/kg/min)
Lipid profile | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean handgrip strenght (pounds)
Session attendance | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean number of program sessions attended
Physical activity | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean minutes per day of objectively measured sedentary, moderate and vigorous physical activity
Waist Circumference | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean waist circumference (cm)
% Fat | 12 months
  Compare changes between the DPP Standard of care group and the DPP+BB intervention group in mean % body fat derived from impedance measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Georgia, Center for Research and Evaluation, Atlanta, Georgia, United States